CLINICAL TRIAL: NCT04625088
Title: Identification of Biometric Marker(s) Capable of Detecting Early Prediabetes: Clinical Trial 1: Antagonism of Hepatic Muscarinic Receptors Attenuates the Postprandial Actions of Hepatic Insulin Sensitizing Substance (HISS)
Brief Title: Identification of Biometric Marker(s) Capable of Detecting Early Prediabetes: Clinical Trial 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SciMar Ltd. (Industry)
Collaborators: Source Nutraceutical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CT-001
Record Dates: First submitted 2020-10-29; First posted 2020-11-12 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Healthy
Keywords: Glucose; Insulin; Prediabetes
MeSH Terms: conditions — Insulin Resistance; Prediabetic State | interventions — Atropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standardized liquid test meal (Experimental)
  Interventions: Other: Standardized liquid test meal
- Atropine + Standardized liquid Test meal (Experimental)
  Interventions: Drug: Atropine + Standardized liquid test meal

INTERVENTIONS:
Other: Standardized liquid test meal — During this study visit, a standardized liquid test meal will be administered. Blood samples will be collected at baseline and then every 30 minutes for 4 hours after test meal.
  Arms: Standardized liquid test meal
Drug: Atropine + Standardized liquid test meal — During this study visit, 1.0 mg atropine will be administered I.V and then a standardized liquid test meal will be administered. Blood samples will be collected at baseline, following atropine administration, and then every 30 minutes for 4 hours after test meal.
  Arms: Atropine + Standardized liquid Test meal

SUMMARY:
The proposed clinical trial is a controlled study of n=24 healthy adult individuals tested in both the Meal-Induced Insulin Sensitization (MIS) state and, following atropine blockade, Absence of Meal-Induced Insulin Sensitization (AMIS) state to differentiate the postprandial glycemia, insulinemia, triglyceride and Hepatic Insulin Sensitizing Substance (HISS) levels in the two states.

The purpose of this study is the identification and development of biometric markers which incorporate the actions and interplay between insulin and HISS. Overall, the study aims to:

1. Utilize a standardized test meal to detect one of the earliest pathologies present during the development of insulin resistance, pre-diabetes and obesity.
2. Compare the control (HISS positive) and post-atropine (HISS negative) tests with the acute consequences of absence of MIS (AMIS) being graphically shown over 4 hours of postprandial nutrient partitioning, tracking the full metabolomic dynamic pattern.
3. To establish values for potential indices (bio-impedance, hand-grip strength, spirometry) in young, fit, lean individuals. These values will be used as baselines for comparative analysis in future clinical trials employing individuals with various degrees of insulin resistance to full Type 2 Diabetes.
4. Demonstrate that these biometric markers can differentiate between the HISS positive and HISS negative post-meal state with the future aim of using the biomarkers for the detection of early prediabetes.

The study will involve 4 study visits: Visit 1 - Prescreening; Visit 2 - Screening; Visit 3 - Liquid test meal administration and postprandial blood collection; Visit 4 - Atropine administration + Liquid test meal administration and postprandial blood collection.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (absence of disease)
* Not on any prescribed medications
* Male and female (in follicular phase)
* 20-40 years of age
* Normal BMI range (18.5-24.9)
* Able to understand and communicate in English
* Comfortable having blood drawn
* Willing to provide urine and blood samples
* Normal urinalysis, Complete Blood Count (CBC) and blood chemistry laboratory test results
* Willingness to undergo bioimpedance testing, handgrip dynamometry (strength) testing, and pulmonary function test (spirometry).
* Willingness to undergo atropine administration
* Willingness to fast for 12 hours prior to the screening and testing days
* Willingness to undergo Electrocardiogram (ECG) and Heart Rate Variability (HRV) testing
* Willingness to use non-hormonal birth control methods throughout the study duration

Exclusion Criteria:

* Glaucoma, Pyloric Stenosis
* Obstructive Uropathy, Urinary Incontinence
* Diabetes, Cardiovascular Disease, including Heart Murmurs
* Diagnosed or with history (last 6 months) and receiving pharma or professional therapy for Psychological/Psychiatric issues
* Inflammatory conditions, including IBD
* Subject on any hormone treatment, including thyroid hormone
* Subject on any steroid therapy including cortisol, or any anti-inflammatory agent
* Sensitivity to anti-cholinergic drugs
* Allergic or have sensitivities to rubbing alcohol during blood draw
* Allergy/sensitivity to any component of the standardized test meal (dextrose, lecithin, soy protein)
* Pregnant women, women of child-bearing potential not willing to use barrier method contraceptives, women trying to get pregnant, and breastfeeding women, women using hormonal birth control
* Whole blood donation (50-499 ml of whole blood) within 30 days, and more than 499 ml of whole blood 56 days prior to test visit 1. Participants should not donate whole blood for the duration of the trial, and for 30 days following the end of the trial
* Blood pressure greater than 140/90 mmHg and heart rate greater than or equal to 80 beats per minute

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
Time course change in serum glucose | Control: Baseline, and every 30 minutes up to 4 hours after test meal administration; Test: Baseline, 15 mins post atropine and every 30 minutes up to 4 hours after test meal administration
  Time course and curve analysis of serum glucose response after the test meal administration with and without atropine pre-treatment.
Time course change in serum insulin | Time Frame: Control: Baseline, and every 30 minutes up to 4 hours after test meal administration; Test: Baseline, 15 mins post atropine and every 30 minutes up to 4 hours after test meal administration
  Time course and curve analysis of serum insulin response after the test meal administration with and without atropine pre-treatment
Time course change in serum triglycerides | Control: Baseline, and every 30 minutes up to 4 hours after test meal administration; Test: Baseline, 15 mins post atropine and every 30 minutes up to 4 hours after test meal administration
  Time course and curve analysis of serum triglycerides response after the test meal administration with and without atropine pre-treatment
Time course change in plasma HISS levels | Time Frame: Control: Baseline, and every 30 minutes up to 4 hours after test meal administration; Test: Baseline, 15 mins post atropine and every 30 minutes up to 4 hours after test meal administration
  Time course and curve analysis of plasma HISS response after the test meal administration with and without atropine pre-treatment

SECONDARY OUTCOMES:
Time course change in serum free fatty acids | Control: Baseline, and every 30 minutes up to 4 hours after test meal administration; Test: Baseline, 15 mins post atropine and every 30 minutes up to 4 hours after test meal administration
  Time course and curve analysis of serum free fatty acid response after the test meal administration with and without atropine pre-treatment
Time course change in plasma lactate | Control: Baseline, and every 30 minutes up to 4 hours after test meal administration; Test: Baseline, 15 mins post atropine and every 30 minutes up to 4 hours after test meal administration
  Time course and curve analysis of plasma lactate response after the test meal administration with and without atropine pre-treatment
Time frame fasted HOMA-IR (Molar Units) | Control: Baseline fasted Test: 15 mins post atropine
  Time frame HOMA-IR, calculated using the formula: fasting insulin (mIU/L) X fasting glucose (mmol/L)
Time course change in Meal Induced Glycemia (MIG) scores (Molar Units) | Control: Every 30 minutes up to 4 hours after test meal administration; Test: Every 30 minutes up to 4 hours after test meal administration
  Time course and curve analysis of Meal Induced Glycemia (MIG) scores response after the test meal administration with and without atropine pre-treatment. MIG is calculated using the formula: MIG = (post meal insulin mIU/L X post meal glucose mmol/L) minus (fasted insulin mIU/L X fasted glucose mmol/L). Higher score equates to a worse (unhealthy) outcome

CONTACTS AND LOCATIONS:
Overall Officials: Vanu Ramprasath, PhD, Principal Investigator — Source Nutraceutical, Inc.
Locations (1):
- Kalo Medical Clinic, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No